CLINICAL TRIAL: NCT00011362
Title: Randomized Clinical Trial of Dexamethasone Therapy in Very-Low-Birth-Weight Infants at Risk for Chronic Lung Disease (CLD)
Brief Title: Dexamethasone Therapy in VLBW Infants at Risk of CLD
Acronym: Dexamethasone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Lu-Ann Papile/ Lead Principal Investigator, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NICHD-NRN-0005; U10HD027881 (NIH); U10HD021373 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD021397 (NIH); U01HD019897 (NIH); U10HD021415 (NIH); U10HD027856 (NIH); U10HD021364 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD027871 (NIH); U10HD021385 (NIH); M01RR000997 (NIH); M01RR008084 (NIH); M01RR000750 (NIH); M01RR000070 (NIH); M01RR006022 (NIH)
Record Dates: First submitted 2001-02-15; First posted 2001-02-19 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Infant, Newborn; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Premature; Bronchopulmonary Dysplasia
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Prematurity; Dexamethasone; Glucocorticoids; Respiratory Distress Syndrome; Respiratory insufficiency; Steroids
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): Dexamethasone
  Interventions: Drug: Dexamethasone Early; Drug: Dexamethasone Late
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Dexamethasone Early; Drug: Dexamethasone Late

INTERVENTIONS:
Drug: Dexamethasone Early — Tapering course of dexamethasone in doses given twice a day (0.25 mg per kilogram of body weight per dose for five days, then 0.15 mg, 0.07 mg, and 0.03 mg per kilogram per dose for three days each), followed by two weeks of saline.
Drug: Dexamethasone Late — Saline for two weeks, followed by either the same tapering two-week course of dexamethasone given to the first group, if the respiratory-index score was >=2.4 on treatment day 14, or an additional two weeks of saline

SUMMARY:
Infants who are on breathing support are often treated with steroids (dexamethasone); however, the best timing of therapy is not known. This trial looked at the benefits and hazards of starting dexamethasone therapy at two weeks of age and four weeks of age in premature infants.

DETAILED DESCRIPTION:
Ventilator-dependent premature infants are often treated with dexamethasone. However, the optimal timing of therapy is unknown. We compared the benefits and hazards of initiating dexamethasone therapy at two weeks of age and at four weeks of age in 371 ventilator-dependent very-low-birth-weight infants (501 to 1500 grams) who had respiratory-index scores (mean airway pressure x the fraction of inspired oxygen) of greater than or equal 2.4 at two weeks of age. The primary outcome was the number of days from randomization to extubation not requiring reintubation (extubation score or death). The secondary outcomes were death before discharge from the hospital; the duration of assisted ventilation, supplementary oxygen therapy and hospital stay; the incidence of chronic lung disease (defined as the need for supplemental oxygen at 36 weeks postconceptional age by best obstetrical estimate) and rates of morbidity and mortality from respiratory causes during the first year. Additional secondary endpoints were hyperglycemia, hypertension, growth, bacteremia, necrotizing enterocolitis and upper GI bleeding.

The sample size of 370 was based on a 0.60 probability that the extubation score of late treatment was greater than early treatment, a 5% two-sided type 1 error, 85% power, and 10% treatment noncompliance.

Infants were randomized to either receive dexamethasone for two weeks followed by saline placebo for two weeks, or saline placebo for two weeks followed by either dexamethasone or additional placebo for two weeks (if they still met entry criteria). Dexamethasone was given at a dose of 0.25 mg per kilogram of body weight twice daily intravenously or orally for five days, and the dose then tapered.

The median time to ventilator independence was 36 days in the dexamethasone-placebo group and 37 days in the placebo-dexamethasone group. The incidences of chronic lung disease (defined as the need for oxygen supplementation at 36 weeks postconceptional age) were 66 percent and 67 percent, respectively. Dexamethasone was associated with an increased incidence of nosocomial bacteremia (relative risk, 1.5; 95 percent confidence interval, 1.1 to 2.1) and hyperglycemia (relative risk, 1.9; 95 percent confidence interval, 1.2 to 3.0) in the dexamethasone-placebo group, elevated blood pressure (relative risk, 2.9; 95 percent confidence interval, 1.2 to 6.9) in the placebo-dexamethasone group, and diminished weight gain and head growth (P less than 0.001) in both groups. Treatment of ventilator-dependent premature infants with dexamethasone at two weeks of age is more hazardous and no more beneficial than treatment at four weeks of age.

ELIGIBILITY:
Inclusion criteria:

* 501 to 1500 grams
* 13 to 15 days old
* Respiratory-index score of greater than or equal to 2.4 that had been increasing or minimally decreasing during the previous 48 hours or a score of greater than or equal to 4.0 even if there had been improvement during the preceding 48 hours

Exclusion criteria:

* Received glucocorticoid treatment after birth
* Had evidence or suspicious signs of sepsis as judged by the treating physician
* Major congenital anomaly of the cardiovascular, pulmonary, or central nervous system

Ages: 13 Days to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 371 (Actual)
Dates: Start 1992-09; Primary Completion 1994-01 (Actual); Study Completion 1994-04 (Actual)

PRIMARY OUTCOMES:
Number of days from randomization to ventilator independence, defined as extubation not requiring reintubation, or extubation followed by elective reintubation for seven days or less so that the infant could undergo a surgical procedure | At hospital discharge

SECONDARY OUTCOMES:
Death before discharge from the hospital | At hospital discharge
Duration of assisted ventilation | At hospital discharge
Duration of supplemental oxygen therapy | At hospital discharge
Duration of hospital stay | At hospital discharge
Incidence of chronic lung disease | At hospital discharge
Morbidity and mortality from respiratory causes during the first year | 12 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Lu-Ann Papile, MD, Principal Investigator — University of New Mexico; Jon E. Tyson, MD MPH, Principal Investigator — University of Texas Southwestern Medical Center; Barbara J. Stoll, MD, Principal Investigator — Emory University; Edward F. Donovan, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Charles R. Bauer, MD, Principal Investigator — University of Miami; Sheldon B. Korones, MD, Principal Investigator — University of Tennessee; James A. Lemons, MD, Principal Investigator — Indiana University School of Medicine; Avroy A. Fanaroff, MD, Principal Investigator — Rainbow Babies & Children's Hospital, Case Western Reserve University; David K. Stevenson, MD, Principal Investigator — Stanford University; Seetha Shankaran, MD, Principal Investigator — Wayne State University; William Oh, MD, Principal Investigator — Women & Infants' Hospital, Brown University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (13):
- United States (13):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - George Washington University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Result] Papile LA, Tyson JE, Stoll BJ, Wright LL, Donovan EF, Bauer CR, Krause-Steinrauf H, Verter J, Korones SB, Lemons JA, Fanaroff AA, Stevenson DK. A multicenter trial of two dexamethasone regimens in ventilator-dependent premature infants. N Engl J Med. 1998 Apr 16;338(16):1112-8. doi: 10.1056/NEJM199804163381604. PMID 9545359
- [Result] Leitch CA, Ahlrichs J, Karn C, Denne SC. Energy expenditure and energy intake during dexamethasone therapy for chronic lung disease. Pediatr Res. 1999 Jul;46(1):109-13. doi: 10.1203/00006450-199907000-00018. PMID 10400143
- [Result] Stoll BJ, Temprosa M, Tyson JE, Papile LA, Wright LL, Bauer CR, Donovan EF, Korones SB, Lemons JA, Fanaroff AA, Stevenson DK, Oh W, Ehrenkranz RA, Shankaran S, Verter J. Dexamethasone therapy increases infection in very low birth weight infants. Pediatrics. 1999 Nov;104(5):e63. doi: 10.1542/peds.104.5.e63. PMID 10545589
- [Result] Lee BH, Stoll BJ, McDonald SA, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Adverse neonatal outcomes associated with antenatal dexamethasone versus antenatal betamethasone. Pediatrics. 2006 May;117(5):1503-10. doi: 10.1542/peds.2005-1749. PMID 16651303
- [Result] Lee BH, Stoll BJ, McDonald SA, Higgins RD; National Institute of Child Health and Human Development Neonatal Research Network. Neurodevelopmental outcomes of extremely low birth weight infants exposed prenatally to dexamethasone versus betamethasone. Pediatrics. 2008 Feb;121(2):289-96. doi: 10.1542/peds.2007-1103. PMID 18245420
- See also: Click here for more information on the NICHD Neonatal Research Network. — http://neonatal.rti.org/